CLINICAL TRIAL: NCT06152978
Title: A Prospective, Open-label, Randomized, Phase II Study of the Efficacy and Safety of Sintilimab Combined With Chemotherapy Versus Chemotherapy in Perioperative Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma (ECTOP-2006).
Brief Title: A Perioperative Sintilimab and Chemotherapy in Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Haiquan Chen, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-2006
Record Dates: First submitted 2022-11-01; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: perioperative; esophageal cancer; programmed cell death protein-1 inhibitor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab plus chemotherapy (Experimental): Sintilimab: 200mg; cisplatin: 75mg/m2, d1, routine hydration for 3 days; nab-paclitaxel: 260mg/m2, d1, every 3 weeks, 2-3 cycles.
  Interventions: Drug: Sintilimab; Drug: Chemotherapy
- Chemotherapy (Active Comparator): Cisplatin: 75mg/m2, d1, routine hydration for 3 days; nab-paclitaxel: 260mg/m2, d1, every 3 weeks, 2-3 cycles.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab (200mg) will be given intravenously on day 1 in 3-week cycles for 2-3 cycles.
  Arms: Sintilimab plus chemotherapy
Drug: Chemotherapy — Cisplatin (75mg/m2) wih routine hydration for 3 days and nab-paclitaxel (260mg/m2) will be given intravenously on day 1 in 3-week cycles for 2-3 cycles.

SUMMARY:
This study is aimed to evaluate the efficacy and safety of sintilimab combined with chemotherapy versus chemotherapy in perioperative treatment of locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study was designed as an open-label, randomized controlled, phase II trial. Subjects will be systematically randomized at a ratio of 1:1 and will be assigned to either the experimental group (sintilimab combined with chemotherapy group) or the control group (chemotherapy alone group). They will receive 2-3 cycles of neoadjuvant therapy followed by radical esophagectomy and lymph node dissection and adjuvant therapy determined by investigators. The primary endpoint is 1-year Event-free survival (EFS) rate.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal squamous cell carcinoma suggested by gastroscopic histopathology.
* The primary tumor is located in the middle and lower of the esophagus.
* cT2-4aN0～3M0 or cT1N+M0 diagnosed by enhanced CT/MRI scan.
* Tumor was evaluated as resectable by surgeon before neoadjuvant therapy.
* Eastern cooperative oncology group (ECOG) performance status of 0 to 1.
* Can eat semi-liquid food.
* Less than 20% body weight loss within 6 months prior to enrollment.
* Sign the consent form before treatment and be able to comply with the relevant procedures such as treatment and visits stipulated in the protocol.
* With adequate organs function 1 week before enrollment and tolerable to chemotherapy and surgery.
* Female subjects of childbearing age or male subjects whose sexual partners are females of childbearing age should take effective contraceptive measures throughout the treatment period and 180 days after the last dose of the test drug.
* Agree and be able to provide archived or fresh pathological tissue and whole blood, urine and fecal samples for biomarker testing.

Exclusion Criteria:

* With metastases or unresectable primary lesion suggested by imaging before treatment.
* History of previous subtotal gastrectomy.
* Patients with active malignancy within 2 years other than the tumor studied in this study or a localized tumor that has been cured such as resected basal or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or breast cancer.
* Received any anti-tumor therapy for the research disease in the past, including radiotherapy, chemotherapy, immunotherapy (including but not limited to interleukin, interferon, thymus hormone) and traditional Chinese medicine therapy.
* With signs of pre-esophageal perforation. With any active autoimmune disease or has a history of autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 12 months
  EFS is defined as the time from R0 resection to disease recurrence or metastases or death for subjects achieving radical resection or the time from enrollment to disease progression or death for subjects not achieving radical resection.

SECONDARY OUTCOMES:
R0 surgery rate | 20 months
  R0 resection is defined as no cancer cells are seen microscopically at the resection margin following surgery.
pCR rate | 20 months
  Pathological Complete Response (pCR) is defined as no viable cancer cells in the hematoxylin and eosin (H&E)-stained slides from the resected tumor and lymph nodes following neoadjuvant treatment.
Disease-free survival (DFS) | 24 months
  DFS is calculated from R0 surgery to the date of recurrence or metastases or death in subjects with radical resection.
Overall Survival (OS) | 24 months
  OS is calculated from the randomization to the date of death from any cause.
adverse events | 24 months
  The incidence of treatment-related adverse events (TRAEs), severe adverse events (SAE), based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No